CLINICAL TRIAL: NCT02061631
Title: Open Label, Non Controlled, Non Randomized, Interventional Study to Evaluate the Response Rate After Induction Therapy With DocEtaxel and CIsplatin in Unresectable Locally Advanced Squamous Cell Carcinoma of heaD and nEck
Brief Title: Study to Evaluate the Response Rate to Therapy With Docetaxel and Cisplatin in Unresectable Locally Advanced Squamous Cell Carcinoma of Head and Neck
Acronym: DECIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCETL06445; U1111-1131-0614 (Other: UTN)
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel, Cisplatin (Experimental): Induction:One-hour intravenous infusion of docetaxel at 75 mg/m2 followed by a 30 minute intravenous infusion of cisplatin at 75 mg/m2. All patients to be pre-medicated with oral dexamethasone at 8 mg twice daily for 3 days, commencing one day before docetaxel infusion. All patients will be premedicated with intravenous dexamethasone 20 mg to be administered before cisplatin infusion. Docetaxel and cisplatin treatments to be repeated every 21 days for three cycles.
  Chemoradiotherapy (CRT): Cisplatin to be administered by 30 minutes intravenous infusion at a dose of 30 mg/m2 weekly starting concomitantly with conventional radiotherapy for a period of 6 weeks. Intravenous cisplatin to be continued for four weeks.
  Radiotherapy: Gross disease dose will be 60 Gy/30 fractions and sub clinical dose 45-50 Gy/30 fractions.
  Interventions: Drug: Cisplatin; Drug: DOCETAXEL XRP6976; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cisplatin — Pharmaceutical form:solution Route of administration: intravenous
Drug: DOCETAXEL XRP6976 — Pharmaceutical form:solution Route of administration: intravenous
Drug: Dexamethasone — Pharmaceutical form:tablet Route of administration: oral
Drug: Dexamethasone — Pharmaceutical form:solution Route of administration: intravenous

SUMMARY:
Primary Objective:

To evaluate the overall response rate (including complete response and partial response) of subjects treated with combination therapy docetaxel and cisplatin followed by the chemoradiotherapy in patients with locally advanced head and neck cancer

Secondary Objective:

To assess the safety and tolerability of combination therapy docetaxel and cisplatin followed by the chemoradiotherapy in patients with locally advanced head and neck cancer

DETAILED DESCRIPTION:
The treatment duration for each patient will be around six months. Patients included in the study will be treated with induction regimen followed by chemo radiotherapy. Within the induction period there are three cycles (Docetaxel + Cisplatin) every 21 days, with follow-up post-induction at day 21 after cycle three. This is followed by chemoradiotherapy consisting of radiotherapy for six weeks and cisplatin every week for four weeks. The post-consolidation follow up is at eight weeks after end of chemoradiotherapy.

ELIGIBILITY:
Inclusion criteria :

* Histologically confirmed, unresectable locally advanced squamous cell carcinoma of head and neck of oral cavity in stage III-IV without evidence of distant metastases.
* No prior chemotherapy or radiation therapy.
* Having at least one measurable lesion in one dimension.
* Age ≥18 and <65 years with Eastern Cooperative Oncology Group ≤ 1.
* Adequate organ function:
* Adequate hematological function
* Adequate hepatic function
* Renal function within normal limits

Exclusion criteria:

* Peripheral neuropathy > grade 1 or other serious diseases (unstable ischaemic heart disease, acute myocardial infarction six months prior to inclusion, history of significant neurological or psychiatric disorder or active peptic ulcer).
* Being treated concomitantly with corticosteroids (except as pre-medication).
* Patients having another type of cancer.
* Previous chemotherapy or radiotherapy.
* Any previous definitive surgery for squamous cell carcinoma of head and neck.
* Severe weight loss (> 20 % of body weight) in the preceding 3 months.
* Hearing loss (> grade 2).
* Pregnancy (pregnancy test result for women of childbearing potential).
* Sexually active females with lack of adequate contraception.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve complete response and partial response according to the Response Evaluation Criteria in Solid Tumors (RECIST) | Day 21 after cycle 3

SECONDARY OUTCOMES:
Proportion of patients who achieve complete response and partial response according to the Response Evaluation Criteria in Solid Tumors (RECIST) | 8 weeks after end of chemoradiotherapy
Number of patients with Adverse Events (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 grade) | From Day 1 cycle 1 up to Day 1 chemoradiotherapy or 30 days after the last cycle of induction therapy, whichever comes first
Number of patients with Adverse Events (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 grade) | From Day 1 chemoradiotherapy up to or 30 days after the last day of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Pakistan, Pakistan